CLINICAL TRIAL: NCT07281014
Title: Unmitigated Aldosterone Signaling During Standard Clinical MRA Dosing
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 2000040063
Record Dates: First submitted 2025-12-03; First posted 2025-12-15 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Heart Failure
Keywords: Spironolactone; Aldosterone
MeSH Terms: conditions — Heart Failure | interventions — Spironolactone; Aldosterone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Placebo/placebo (Placebo Comparator): This study will employ a randomized placebo-controlled, double-blind, double-dummy, crossover design testing combinations
  1) IV Vehicle infusion plus oral placebo pill 2) IV Vehicle infusion plus oral 25mg spironolactone 3) IV Aldosterone infusion plus oral placebo pill 4) IV Aldosterone infusion plus oral 25 mg spironolactone on Day 14, 29, 44, 59.
  Interventions: Drug: Placebo
- Placebo/Sprironolactone (Active Comparator): This study will employ a randomized placebo-controlled, double-blind, double-dummy, crossover design testing combinations
  1) IV Vehicle infusion plus oral placebo pill 2) IV Vehicle infusion plus oral 25mg spironolactone 3) IV Aldosterone infusion plus oral placebo pill 4) IV Aldosterone infusion plus oral 25 mg spironolactone on Day 14, 29, 44, 59.
  Interventions: Drug: Placebo; Drug: Spironolactone 25mg
- placebo/aldosterone (Active Comparator): This study will employ a randomized placebo-controlled, double-blind, double-dummy, crossover design testing combinations
  1) IV Vehicle infusion plus oral placebo pill 2) IV Vehicle infusion plus oral 25mg spironolactone 3) IV Aldosterone infusion plus oral placebo pill 4) IV Aldosterone infusion plus oral 25 mg spironolactone on Day 14, 29, 44, 59.
  Interventions: Drug: Placebo; Drug: Aldosterone
- aldosterone/spironolactone (Active Comparator): This study will employ a randomized placebo-controlled, double-blind, double-dummy, crossover design testing combinations
  1) IV Vehicle infusion plus oral placebo pill 2) IV Vehicle infusion plus oral 25mg spironolactone 3) IV Aldosterone infusion plus oral placebo pill 4) IV Aldosterone infusion plus oral 25 mg spironolactone on Day 14, 29, 44, 59.
  Interventions: Drug: Spironolactone 25mg; Drug: Aldosterone

INTERVENTIONS:
Drug: Placebo — This study will employ a randomized placebo-controlled, double-blind, double-dummy, crossover design testing combinations
  1) IV Vehicle infusion plus oral placebo pill 2) IV Vehicle infusion plus oral 25mg spironolactone 3) IV Aldosterone infusion plus oral placebo pill 4) IV Aldosterone infusion plus oral 25 mg spironolactone on Day 14, 29, 44, 59.
  Arms: Placebo/Sprironolactone; Placebo/placebo; placebo/aldosterone
Drug: Spironolactone 25mg — This study will employ a randomized placebo-controlled, double-blind, double-dummy, crossover design testing combinations
  1) IV Vehicle infusion plus oral placebo pill 2) IV Vehicle infusion plus oral 25mg spironolactone 3) IV Aldosterone infusion plus oral placebo pill 4) IV Aldosterone infusion plus oral 25 mg spironolactone on Day 14, 29, 44, 59.
  Arms: Placebo/Sprironolactone; aldosterone/spironolactone
Drug: Aldosterone — This study will employ a randomized placebo-controlled, double-blind, double-dummy, crossover design testing combinations
  1) IV Vehicle infusion plus oral placebo pill 2) IV Vehicle infusion plus oral 25mg spironolactone 3) IV Aldosterone infusion plus oral placebo pill 4) IV Aldosterone infusion plus oral 25 mg spironolactone on Day 14, 29, 44, 59.
  Arms: aldosterone/spironolactone; placebo/aldosterone

SUMMARY:
The purpose of this research study is to understand the biology related to the potential shortcomings of existing anti-aldosterone therapy.

DETAILED DESCRIPTION:
This is a randomized, double blind, double dummy, placebo-controlled, crossover study where aldosterone will be infused intravenously (IV) with and without guideline recommended low dose oral mineralocorticoid receptor antagonists therapy. Participants will receive, in a randomized order, 1) IV Vehicle infusion plus oral placebo pill 2) IV Vehicle infusion plus oral 25mg spironolactone 3) IV Aldosterone infusion plus oral placebo pill 4) IV Aldosterone infusion plus oral 25 mg spironolactone. Each crossover period will be separated by 2 weeks to allow for steady state blood level of spironolactone and metabolites to be reached (or complete washout from prior spironolactone). The broad study design will be designed around evaluation of change in urine sodium to potassium ratio, sodium output following a sodium chloride challenge, and collecting the necessary biospecimens to test our hypotheses.

ELIGIBILITY:
Inclusion Criteria:

1. Chronic stable heart failure at optimal volume status. Inclusion will require participants to be NYHA class I or II.
2. eGFR > 30 ml/min/1.73m2
3. Serum potassium ≤5.0 meq/L and ≥3.5 meq/L
4. Stable heart failure medications without need or expectation for changes during the 8-week study period
5. Free from heart failure decompensation for the preceding 60 day
6. Systolic blood pressure >90 mmHg if not taking an MRA at screening. If patients are already taking an MRA at the time of screening a systolic blood pressure needs to be >80 mmHg.

Exclusion Criteria:

1. Uncontrolled hypertension (SBP > 160 mmHg)
2. Severe bladder dysfunction
3. Current MRA dose > 50mg spironolactone or equivalent or non MRA potassium sparing diuretic such as amiloride
4. Contraindication to initiation or withdrawal of spironolactone per study procedures
5. History of severe hyperkalemia (K>6.0 meq/l)
6. Brittle volume sensitive heart failure, recurrent flash pulmonary edema, restrictive cardiomyopathy or other pathology that would make aldosterone infusion high risk
7. Pregnant or breastfeeding
8. Women of childbearing potential that are not receiving a highly effective form of contraception. Females of childbearing potential must agree to use a highly effective method of birth control until 14 days after the last dose of study drug. The following are highly effective methods for this study:

   * Combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation: oral, intravaginal, or transdermal
   * Progestogen-only hormonal contraception associated with inhibition of ovulation: oral, injectable, or implantable
   * Intrauterine device (IUD)
   * Intrauterine hormone-releasing system (IUS)
   * Bilateral tubal occlusion
   * Vasectomized partner
   * Sexual abstinence

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
change in urine sodium to potassium ratio | 59 days
  Change in sodium to potassium ratio between aldosterone vs vehicle infusion during the spironolactone vs. placebo arms.

SECONDARY OUTCOMES:
Urine Sodium output following saline load | 59 days
  Effect of MRA and aldosterone infusion on natriuresis following a saline load
Natriuretic effect of adjuvant to loop diuretic therapy | 59 days
  Effect of MRA and aldosterone infusion on natriuresis following IV bumetanide challenge

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Testani, MD, Principal Investigator — Yale University
Locations (1):
- Yale University, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No